CLINICAL TRIAL: NCT05411978
Title: A Multi-center, Randomized, Double-blind, Placebo-controlled Parallel Pilot Study to Evaluate Safety and Efficacy of Oral Idebenone for Preventive Treatment of Migraine in Adult Migraine Patients
Brief Title: Safety and Efficacy of Oral Idebenone for Preventive Treatment of Migraine in Adult Migraine Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Yonggang.wang, Director, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ADBK-3101-303-002
Record Dates: First submitted 2022-05-31; First posted 2022-06-09 (Actual); Last update posted 2022-06-23 (Actual); Status verified 2022-06

CONDITIONS: Migraine
Keywords: Migraine Prophylaxis; Mitochondrial Dysfunction; Idebenone Individualized Treatment
MeSH Terms: conditions — Migraine Disorders; Mitochondrial Diseases | interventions — idebenone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Idebenone 30 mg+ Placebo 60 mg (Placebo Comparator): Idebenone 30 mg+ placebo 60 mg TID Oral ,for 12 weeks
  Interventions: Drug: Idebenone+ placebo
- Idebenone 90 mg (Experimental): Idebenone 90 mg TID Oral ,for 12 weeks
  Interventions: Drug: Idebenone
- Placebo 90 mg (Placebo Comparator): Placebo 90 mg TID Oral,for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Idebenone+ placebo — Participants will receive Idebenone 30 mg+ placebo 60 mg for 12 weeks.
  Other Names: Idebenone 30 mg+ placebo 60 mg
  Arms: Idebenone 30 mg+ Placebo 60 mg
Drug: Idebenone — Participants will receive Idebenone 90 mg for 12 weeks.
  Other Names: Idebenone 90 mg
  Arms: Idebenone 90 mg
Drug: Placebo — Participants will receive Placebo 90 mg for 12 weeks
  Other Names: Placebo 90 mg
  Arms: Placebo 90 mg

SUMMARY:
This is a multi-center, prospective, double-blind randomized controlled trial on a sample of patients with migraine. Subjects will only be enrolled when a physician or research assistant who is familiar with the study protocol is available to enroll patients. Written, informed consent will be obtained from each patient. Consent will include a discussion of the risks and benefits.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants ages 18 to 65 years;
* At least a 1-year history of migraine with or without aura is consistent with a diagnosis according to the ICHD-3;
* Migraine onset before age 50 years;
* History of 4 to 15 migraine attacks days per month in each of the 3 months prior to the screening visit;
* The number of headache attacks <15 days/month during the 3 months prior to the screening visit;
* Be willing to use effective contraception during the trial and for 28 days after the end of the last dose;
* Sign the informed consent form.
* History of 4 to 14 migraine attacks days within 4 weeks during the screening visit.
* The number of headache attacks <14 days/month within 4 weeks during the screening visit;
* Completed at least 23 days of the electronic diary within 28 days during the screening visit. And the participant is to be able to read, understand and complete the study questionnaire and headache diary;
* Understand and comply with the study procedures and methods, and voluntarily participate in this study.

Exclusion Criteria:

* Participants diagnosed with probable migraine by ICHD-3
* Current or previous diagnosis of primary, secondary, or painful cranial neuropathy other than migraine (diagnostic criteria according to ICHD-3)
* Prior ineffectiveness after adequate treatment with more than 2 medications, which are listed below: Divalproex, sodium valproate; topiramate; beta-blockers; Tricyclic antidepressants; serotonin-norepinephrine reuptake inhibitors; Flunarizine, Verapamil; Lisinopril, Candesartan.

Definition of failure to treat: frequency, duration, and severity of headache 6 weeks after administration of the degree of the above drug does not decrease.

* Use of other devices or prohibited medications such as painkillers containing opioids for the treatment of migraine within 2 months before or during the screening visit
* Therapeutic injections of Botulinum toxin in the head, face, or neck within 4 months before screening and during the study periods
* Simultaneous use of 2 or more drugs within 2 months before or during the screening visit may be prophylactic Medications for migraine effects (if used only 1 prophylactic drug, the dose must be stable for 2 months before the screening visit and throughout the study period)
* The following situations occur within 2 months before the screening period begins: take ergotamines or triptans at least 10 days per month, or take non-steroidal anti-inflammatory drugs (NSAID) only every month ≥15 days, NSAID combination ≥10 days, or use opioid or barbiturate analgesics ≥4 days per month;
* Participants use the prohibited drugs such as painkillers containing opioids, devices, or regimens during treatment.
* History of active chronic pain syndrome (e.g., fibromyalgia, chronic pelvic pain, face Pain, etc.);
* History of mental illness (e.g., schizophrenia or bipolar disorder) or Patient Health Questionnaire (PHQ-9) score ≥15. If the participant has a history of anxiety or depression (PHQ-9 score < 15) and takes no more than one psychotropic drug, the participant will be allowed to enter. (participant must take a steady dose of treatment within 3 months before the screening visit)
* Severe neurological disorders other than migraines (including febrile seizures);
* History of a malignant tumor within 5 years before the screening visit, except for non-melanoma skin cancer, cervical or ductal carcinoma in situ;
* The screening visit meets any of the following laboratory test values: Alanine transaminase (ALT) or aspartate aminotransferase(AST) >1.5×ULN, or total bilirubin >1.5×ULN (except for participants diagnosed with Gilbert syndrome);
* History of myocardial infarction, stroke, or transient ischemic attack, unstable angina or coronary bypass surgery within 12 months before the screening visit
* Expose participants to significant risk or confuse the study
* Based on clinical interviews or C-SSRS, the investigator believes that the subject has self-harmed or harmed him Human risk;
* History of drugs or alcohol abuse within 12 months before the screening visit
* Pregnant, planning pregnancy, or Lactating women;
* Fertile female participants are unwilling to use an effective contraceptive during the study period Method.

Infertile women as follows: history of menopause, age ≥ 55 years, menopause ≥12 months.

Age < 55 years, free from spontaneous menstruation for at least 2 years. Age < 55, has spontaneous menstruation in the past 1 year, but currently amenorrhea (e.g., Spontaneous or secondary to hysterectomy), and postmenopausal gonadotropin levels gonadotropin Luteinizing hormone (LH), follicle-stimulating Hormone> 40 IU/L or postmenopausal estradiol level <5 ng/dL History of bilateral oophorectomy, hysterectomy, or bilateral salpingectomy

* Participated in other clinical trials within the first 3 months
* Known allergy to Idebenone or any of its ingredients(e.g., lactose intolerant)；
* The participants are employees or immediate family members of the research center (parents, spouses, siblings, or children).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2022-05-09 (Actual); Primary Completion 2024-06-20 (Estimated); Study Completion 2024-06-20 (Estimated)

PRIMARY OUTCOMES:
Changes in the migraine days per 4 weeks relative to the baseline. | baseline, 4,8,12 weeks
  Days with migraine in the last four weeks from a daily headache diary.

SECONDARY OUTCOMES:
Frequency of headache attacks per 4 weeks as compared to baseline. | baseline,at 4,8,12 weeks
  Headache attack as any consistent headache attacks or the use of specific headache drugs.
Changes in the moderate / severe headache days per 4 weeks relative to the baseline | baseline,at 4,8,12 weeks
  Moderate / severe headache days as a day in which moderate or severe pain persists for at least 4 hours, or headache lasts for one day after successful medication for acute headache.
Percentage of participants with at Least 50%, 75% and 100% reduction in the Number of Days of Migraine Attacks per 4 weeks. | baseline,at 4,8,12 weeks
  The response rate as the percentage reduction in the frequency of migraine attacks (or days of migraine, or days of moderate or severe headache) compared with the baseline during each treatment period.
Change in frequency of acute drug use per 4 weeks relative to baseline. | baseline,at 4,8,12 weeks
  The allowed medications include the following categories of drugs: triptans, ergots, opioids, analgesics (including acetaminophen), NSAIDs (including aspirin), and antiemetics.
Change in dose of acute drug use per 4 weeks relative to baseline. | baseline,at 4,8,12 weeks
  The allowed medications include the following categories of drugs: triptans, ergots, opioids, analgesics (including acetaminophen), NSAIDs (including aspirin), and antiemetics.
Change in peak headache pain intensity per 4 weeks relative to baseline. | baseline,at 4,8,12 weeks
  Participates record the maximum intensity of daily headaches and any medication used. The Visual Analogue Scale (VAS) can be used instead of or in conjunction with a 4-level classified rating scale.
Change in average headache intensity per 4 weeks relative to baseline. | baseline,at 4,8,12 weeks
  Four-point rating scale to evaluate the headache intensity of each migraine day--painless, mild, moderate, or severe. The Visual Analogue Scale (VAS) can be used instead of or in conjunction with a 4-level classified rating scale.
Change in cumulative hours of moderate/severe headache pain per 4 weeks relative to baseline. | baseline,at 4,8,12 weeks
  The cumulative number of hours of moderate / severe pain calculated by electronic headache diaries. If an attack occurs before going to bed and when you wake up, the amount of sleep also counts as the number of headache hours.
Change in the number of without symptoms days per 4 weeks relative to baseline. | baseline,at 4,8,12 weeks
  The number of days without aura, prodromal symptoms, headaches, pain, and subsequent symptoms by headache diary.
Change in the number of without headache days per 4 weeks relative to baseline. | baseline,at 4,8,12 weeks
  The number of days without headaches by headache diary.
Change in The Fatigue Severity Scale (FSS) score per 4 weeks relative to baseline. | baseline,at 4,8,12 weeks
  The Fatigue Severity Scale (FSS) is a method of evaluating the impact of fatigue on you. The FSS is a short questionnaire that requires you to rate your level of fatigue. The FSS questionnaire contains nine statements that rate the severity of your fatigue symptoms. Read each statement and circle a number from 1 to 7, based on how accurately it reflects your condition during the past week and the extent to which you agree or disagree that the statement applies to you. A higher score indicates greater severity.
Change in The Modified Migraine Disability Assessment Scale score per 4 weeks relative to baseline. | baseline,at 4,8,12 weeks
  The Modified Migraine Disability Assessment Scale is a 7-item questionnaire designed. The score is the sum of missed work or school days, days at work or school plus days of household work where productivity was reduced by half or more, missed household work days, and missed non-work activity days due to headaches in the last 1 months.
Change in The Headache Impact Test(HIT-6) score per 4 weeks relative to baseline. | baseline,at 4,8,12 weeks
  The HIT-6 is a 6-question assessment used to measure the impact headaches have on a participant's ability to function on the job, at school, at home, and in social situations. It assesses the effect that headaches have on normal daily life and the participant's ability to function.
  Responses are based on frequency using a 5-point scale ranging from "never" to "always." The HIT-6 total score, which ranges from 36 to 78, is the sum of the responses - each of which is assigned a score ranging from 6 points (never) to 13 points (always).
Change in The Migraine-Specific Quality-of-Life Questionnaire, Version 2.1 (MSQ Version 2.1) score per 4 weeks relative to baseline. | baseline,at 4,8,12 weeks
  The MSQ v2.1 is a 14-item questionnaire designed to measure health-related quality-of-life impairments attributed to migraine in the past 4 weeks. It is divided into 3 domains: Role Function Restrictive assesses how migraines limit one's daily social and work-related activities; Role Function Preventive assesses how migraines prevent these activities; and the Emotional Function domain assesses the emotions associated with migraines.
Patient Global Impression of Change (PGIC). | baseline,at 4,8,12 weeks
  The PGIC is a single item questionnaire used to measure the participant's impression of overall change in migraine since the first dose of study medication. The measure uses a 7-point rating scale with responses ranging from "very much better" to "very much worse."
Change in The Patient Health Questionnaire-9 (PHQ-9) score per 4 weeks relative to baseline. | baseline,at 4,8,12 weeks
  The PHQ-9 is the depression module, which scores each of the 9 DSM-IV criteria as "0" (not at all) to "3" (nearly every day). A PHQ-9 score total of 0-4 points equals "normal" or minimal depression. Scoring between 5-9 points indicates mild depression, 10-14 points indicates moderate depression, 15-19 points indicates moderately severe depression, and 20 or more points indicates severe depression.
Change in The General Anxiety Disorder-7(GAD-7) score per 4 weeks relative to baseline. | baseline,at 4,8,12 weeks
  GAD-7 is a proven, self-administered and concise tool for screening and diagnosing mental health disorders, which has been tested in the field in office practice. The GAD-7 scale score ranges from 0 to 21.
Change in The Functional Impairment Scale (FIS) score per 4 weeks relative to baseline. | baseline,at 4,8,12 weeks
  Functional impairment scale (FIS) is a 4-point scale to evaluate the functional status and injury intensity in daily activities. It can be used in conjunction with the four-point pain intensity scale, usually done daily and summarized within four weeks.
Change in The European Quality of Life 5 Dimensions 3 Level Version (EQ-5D-3L) scores per 4 weeks relative to baseline. | baseline,at 4,8,12 weeks
  EQ-5D-3L is a generic instrument for use as a measure of health status. The EQ-5D-3L consists of 2 components-the EQ-5D descriptive system and the EQ VAS. The descriptive system comprises of 5 dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression). The respondent is asked to indicate his/her health state by ticking (or placing a cross) in the box against the most appropriate statement in each of the 5 dimensions.
  The EQ VAS records the respondent's self-rated health on a vertical, VAS where the endpoints are labelled "Best imaginable health state" and "Worst imaginable health state." The scoring range of the EQ VAS is from 0 (worst imaginable health) to 100 (best imaginable health).
Change in The Columbia-Suicide Severity Rating Scale (C-SSRS) score per 4 weeks relative to baseline. | baseline,at 4,8,12 weeks
  C-SSRS will be administered to study subjects at each study visit to assess possible suicidal ideation and behavior. Reports of suicidal ideation with intent to act (endorse item 4 or 5) and reports of actual, aborted, or interrupted suicide attempts or a behavior preparatory for making an attempt indicate subjects at high risk for suicide.

CONTACTS AND LOCATIONS:
Locations (1):
- Yonggang Wang, Beijing, China